CLINICAL TRIAL: NCT03663465
Title: The Disparity of Hawthorn Effects to Triglyceride/High-density Lipoprotein Cholesterol Ratio in Schizophrenics With Antipsychotics
Brief Title: The Effect of Hawthorn on Lipoprotein Cholesterol Ratio in Schizophrenics With Antipsychotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calo Psychiatric Center (Other)
Responsible Party: Principal Investigator, For-Wey Lung, Superintendent and Attending physician, Calo Psychiatric Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MAB101-109
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Schizophrenia
Keywords: Hawthorn; TG/HDL ratio; dyslipidemia; schizophrenia; antipsychotics
MeSH Terms: conditions — Schizophrenia; Dyslipidemias | interventions — crataegus extract

STUDY DESIGN:
Intervention Model Description: case control study
Who Masked: Participant, Investigator
Masking Description: two groups of participants and investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hawthorn and SGAs (Experimental): SGAs has a dose of 3-20 gm/day, Hawthorn at a dose of 3 gm/day for six months.
  Interventions: Other: Hawthorn; Drug: SGAs
- Hawthorn (Active Comparator): Hawthorn at a dose of 3 gm/day for six months.
  Interventions: Other: Hawthorn

INTERVENTIONS:
Other: Hawthorn — Hawthorn tablet
Drug: SGAs — SGAs tablet
  Other Names: second-generation antipsychotics
  Arms: Hawthorn and SGAs

SUMMARY:
Importance: The problems of side effects of metabolic disturbances in schizophrenic patients have been of worldwide concern for some time. Patients with dyslipidemia have an increased risk of cardiovascular diseases. A Chinese herb, Hawthorn, is widely used for the treatment of dyslipidemia.

Objective: Therefore, this study aimed to investigate the effect of Hawthorn on lipid profile levels in schizophrenic patients treated with antipsychotics.

Design, Setting, and Participants: A longitudinal case-control study was used in a general hospital in Taiwan. A total of 59 schizophrenics treated with antipsychotics, and 76 healthy adult subjects, who were all hospital workers, were enrolled in this study.

Main outcomes and measures: All participants received Hawthorn at a dose of 3 gm/day for six months.

DETAILED DESCRIPTION:
The problem of metabolic disturbances in schizophrenic patients who take antipsychotics has always been a cause for global concern and discussion. Although Hawthorn is widely used in the treatment of heart problems and the lowering of blood lipid levels, it is unknown whether Hawthorn has an effect in schizophrenic patients treated with antipsychotics. Hence, there are several areas of interest in the present study: 1) the effect of Hawthorn on lipid profile levels in schizophrenic patients treated with antipsychotics; 2) a comparison of lipid profile levels between schizophrenic patients and healthy adults; 3) the contributing factors that relate to changes in lipid profile levels in patients who take Hawthorn.

ELIGIBILITY:
Inclusion Criteria:

* Patients in case group who had to meet the diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
* All participants in the case group had previously received antipsychotic treatment for a period of time.

Exclusion Criteria:

* Patients who had comorbid serious medical illnesses, and may therefore present substantial clinical risk due to pharmacotherapy, were excluded from the sample
* Participants were pregnant and lactating women in both group, were excluded.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
lipid profiles | three days
  lipid profiles (including TC, TG, HDL, LDL) were collected three times (at first week, 12th week and 24th week. Total collecting day were three days.